CLINICAL TRIAL: NCT03406611
Title: A Double Blind, Randomized, Placebo-controlled, Phase 1/2 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Effects on Clinical Outcomes of Pegtibatinase (TVT-058), Administered Subcutaneously in Patients with Cystathionine Beta-Synthase Deficient Homocystinuria (COMPOSE)
Brief Title: Pegtibatinase As an Enzyme Therapy for Patients with Homocystinuria Caused by Cystathionine Beta-Synthase Deficiency (COMPOSE)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBS-HCY-CT-01
Record Dates: First submitted 2017-12-05; First posted 2018-01-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pegtibatinase (Active Comparator)
  Interventions: Drug: Pegtibatinase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pegtibatinase — Pegtibatinase sterile solution for subcutaneous injection
  Other Names: TVT-058; OT-58; PEG modified CBS, PEG htCBS C15S, htCBS C15S ME-200GS
  Arms: Pegtibatinase
Drug: Placebo — Normal saline for subcutaneous injection
  Arms: Placebo

SUMMARY:
Homocystinuria caused by Cystathionine Beta-Synthase (CBS) Deficiency is a rare autosomal-recessive metabolic condition characterized by an excess of homocysteine (Hcy) in the plasma, tissues and urine. It is due to reduced or absent activity of the CBS enzyme, and is also known as classical homocystinuria. The symptoms associated with homocystinuria are variable in severity and time of onset across patients. Some affected individuals may have mild signs of the disorder; others may have multi-systemic involvement including potentially life-threatening complications. Homocystinuria can affect many different organ systems of the body; the four most commonly involved are the eyes, central nervous system, skeleton, and the vascular system.

The current approaches to treatment of homocystinuria patients include a highly restrictive diet and use of dietary supplements. Lifetime compliance with this diet is poor. Pegtibatinase (TVT-058) represents a novel therapeutic approach that incorporates the use of a modified version of the native, human CBS (hCBS) enzyme. The goal of treatment is to introduce the CBS enzyme into circulation, resulting in reduced Hcy levels, increased cystathionine (Cth) and cysteine (Cys) levels.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of homocystinuria based on genetic confirmation and plasma tHcy ≥50 micromoles and documentation of previous tHcy level ≥80 micromoles
* Willing and able to provide written, signed informed consent and to comply with all study related procedures.
* Subjects born biologically as female who are of child-bearing potential must have a negative pregnancy test at screening and be willing to have additional pregnancy tests during the study. Subjects born biologically as male who identify as female and are not of childbearing potential are not required to undergo pregnancy tests
* Sexually active subjects who have childbearing potential or those who have partners of childbearing potential must be willing to use acceptable methods of contraception while on the study and for 4 weeks after the end of study
* Willing to maintain a stable diet with no significant modifications while on study and complete a daily diet diary.

Exclusion Criteria:

* Previous exposure to pegtibatinase and/or previous participation in a clinical trial that included administration of pegtibatinase
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or while on study
* Use or planned use of any injectable drugs containing PEG (other than pegtibatinase or COVID-19 vaccines), including medroxyprogesterone (eg, Depo-Provera) injection, within 3 months prior to Screening and during study participation
* Known hypersensitivity to PEG-containing product or any components of pegtibatinase
* A positive test for HIV antibody, hepatitis B surface antigen, or hepatitis C antibody
* A history of organ transplantation, chronic immunosuppressive therapy, or substance abuse
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study
* Concurrent disease or condition or planned major surgery that would interfere with study participation or safety in the opinion of the investigator.
* Any condition that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study
* Major surgery planned during the study period

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | Through double-blind study completion, approximately 10 months per patient
  Incidence of AEs (by type, severity and relationship to study drug)
Anti-pegtibatinase antibodies | Through double-blind study completion, approximately 10 months per patient
  Presence and levels of anti-pegtibatinase antibodies in plasma as measured by antibody titers
Anti-PEG antibodies | Through double-blind study completion, approximately 10 months per patient
  Presence and levels of anti-PEG antibodies in plasma as measured by antibody titers

SECONDARY OUTCOMES:
Changes in pegtibatinase levels | Through double-blind study completion, approximately 10 months per patient
  Changes in pegtibatinase levels following single and repeat administration at specified timepoints
Changes in Met cycle metabolites levels - tHcy | Through double-blind study completion, approximately 10 months per patient
  Changes in total homocysteine levels in micromoles
Changes in Met cycle metabolites levels - total Cys | Through double-blind study completion, approximately 10 months per patient
  Changes in total cysteine levels in micromoles
Changes in Met cycle metabolites levels - Met | Through double-blind study completion, approximately 10 months per patient
  Changes in methionine levels in micromoles
Changes in Met cycle metabolites levels - Cth | Through double-blind study completion, approximately 10 months per patient
  Changes in cystathionine levels in micromoles
Changes in Met cycle metabolites levels - Phe | Through double-blind study completion, approximately 10 months per patient
  Changes in phenylalanine levels in micromoles
Descriptive ophthalmology examination findings | Through double-blind study completion, approximately 10 months per patient
  Comprehensive ophthalmological examination (for each eye: visual acuity [myopia, hyperopia, exotropia], slit lamp examination [ectopic lentis, cataracts, corneal abrasion, and uveitis], retinal examination [retinal degeneration, retinal detachment, retinitis pigmentosa, uveitis)]). Assessment of presence and severity of findings.
Bone densitometry using dual-energy X-ray absorptionmetry (DEXA) scans | Through double-blind study completion, approximately 10 months per patient
Cognitive assessments using the National Institutes of Health Toolbox Cognition Battery score | Through double-blind study completion, approximately 10 months per patient
Patient Reported Outcome (PRO): Quality of Life in Neurological Disorders [Neuro-QoL] | Through double-blind study completion, approximately 10 months per patient
  The Quality of Life in Neurological Disorders [Neuro-QoL] includes Anxiety Short Form, Depression Short Form, Satisfaction with Social Roles Short Form, Cognition Function Short Form for 18+ years of age; Anxiety Short Form, Depression Short Form, Social Relations - Interaction with Peers Short Form, and Cognitive Function Short Form for Ages 12 to 17 years old
Patient Reported Outcome (PRO): Quality of Life by 36-Item Short Form Survey [SF-36] | Through double-blind study completion, approximately 10 months per patient
Patient Reported Outcome (PRO): Quality of Life by EuroQol 5-Dimentional Instrument [EQ 5D] | Through double-blind study completion, approximately 10 months per patient

CONTACTS AND LOCATIONS:
Overall Officials: Michael Imperiale, MD, Study Director — Travere Therapeutics, Inc.
Locations (8):
- United States (8):
  - Travere Investigational Site - Virtual Site, Culver City, California
  - Travere Investigational Site, Aurora, Colorado
  - Travere Investigational Site, Miami, Florida
  - Travere Investigational Site, Indianapolis, Indiana
  - Travere Investigational Site, Portland, Maine
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.